CLINICAL TRIAL: NCT06817278
Title: Internet-delivered Emotion Regulation Individual Therapy or Adolescents (IERITA) With Self-injury Within Child and Adolescent Mental Health Services: Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Region Skane (Other); Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Olivia Ojala, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-01916
Record Dates: First submitted 2025-01-16; First posted 2025-02-10 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-01

CONDITIONS: Nonsuicidal Self-Injury; Self-Harm
Keywords: Nonsuicidal self-injury; Internet-delivered treatment; Self-harm; Adolescence
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be masked to allocation and classification. Therapists will be masked until treatment week four.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptable Internet-delivered emotion regulation individual therapy adjunctive to treatment as usual (Experimental): Participants will receive Internet-delivered Emotion Regulation Individual Therapy (IERITA) for 12 weeks. Adolescents allocated to experimental arm and classified as likely non-remission, will change to adapted IERITA in treatment week four. Adolescents allocated to experimental arm and classified as likely remission will continue standard IERITA. In addition to IERITA, participants are free to will receive any type of treatment as usual for 12 weeks as provided in the community.
  Interventions: Behavioral: Adaptable IERITA; Other: Treatment as usual
- Standard Internet-delivered emotion regulation individual therapy adjunctive to treatment as usual (Active Comparator): Participants will receive Internet-delivered Emotion Regulation Individual Therapy (IERITA) for 12 weeks. All participants will continue standard IERITA throughout the treatment period. In addition to IERITA, participants are free to will receive any type of treatment as usual for 12 weeks as provided in the community.
  Interventions: Behavioral: Standard IERITA; Other: Treatment as usual

INTERVENTIONS:
Behavioral: Adaptable IERITA — IERITA is a 12-week acceptance-based behavioral therapy. The goal is to reduce self-injury through learning and using other ways to regulate emotions. IERITA includes modules where the participants can read text, watch videos, listen to audio, and message their allocated therapists. The adolescent treatment is 11 modules, and the parent course is six. Both adolescents and parents receive separate asynchronous online therapist support. The adapted IERITA intervention is tailored to the participant and can thus entail different adaptions for different participants. Adaptions can entail changes in therapist contact, what material to focus on, and how to work with the treatment. The adapted IERITA intervention is offered between week four and 12.
  Arms: Adaptable Internet-delivered emotion regulation individual therapy adjunctive to treatment as usual
Behavioral: Standard IERITA — IERITA is a 12-week acceptance-based behavioral therapy. The goal is to reduce self-injury through learning and using other ways to regulate emotions. IERITA includes modules where the participants can read text, watch videos, listen to audio, and message their allocated therapists. The adolescent treatment is 11 modules, and the parent course is six. Both adolescents and parents receive separate asynchronous online therapist support.
  Arms: Standard Internet-delivered emotion regulation individual therapy adjunctive to treatment as usual
Other: Treatment as usual — Participants are free to any receive regular care (i.e., psychosocial treatment, medications, or a combination of both) as needed during the trial.

SUMMARY:
The overall purpose of the study is to implement and evaluate IERITA (Internet-delivered Emotion Regulation Individual Therapy for Adolescents) within child and adolescent mental health services for adolescents engaging in nonsuicidal self-injury (NSSI) and to optimize treatment outcomes for those adolescents at risk of insufficient effects. The specific purpose of this pilot trial is to investigate feasibility in preparation for a larger trial.

DETAILED DESCRIPTION:
Self-injury without the intention to die is a growing and urgent global health crisis among youth. It is associated with substantial individual and societal costs, including increased risk of suicide attempts. Scalable and evidence-based treatments are needed but lacking. Digital interventions can be one promising solution. A recent study shows that a novel brief digital treatment, IERITA, can be efficacious compared to treatment as usual only. However, not all respond sufficiently to standardized treatment, such as IERITA, and continued self-injury entails risks and suffering.

In this randomized controlled pilot trial, participants will be randomly allocated (1:1) to standard IERITA or adaptable IERITA. All participants will first receive standard IERITA for four weeks. In treatment week four, non-remission will be predicted. Adolescents allocated to adaptable IERITA and classified as likely non-remission, will change to adapted IERITA for the remaining eight weeks while all other participants will continue standard IERITA. Data will be collected pre-treatment, during treatment, post-treatment, one- three- and twelve-month post-treatment. The primary endpoint is one-month post-treatment.

The main objective is to investigate the project's feasibility and test key components. The specific objectives are:

1. Examine the feasibility of the project (treatment satisfaction and adherence, degree of participation in data collection, and level of resources).
2. Explore the utility of adapted IERITA compared to standard IERITA for adolescents at risk of non-remission.
3. Evaluate the performance of the algorithm predicting treatment non-remission.

This project is sponsored by the Swedish Research Council for Health, Working life, and Welfare (number 2024-01916)

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years old
* At least one self-injury episode in the past three months
* A parent willing to engage in the parent program

Exclusion Criteria:

* Immediate suicide risk
* Global functioning corresponding to a rating ≤40 of the Children's Global Assessment Scale (CGAS)
* Social problems needing immediate intervention (e.g., violence within the family)
* Ongoing dialectical behavior therapy for adolescents

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Deliberate Self-harm Inventory - Youth version (DSHI-Y) | One-, three- and twelve-months post-treatment
  The DSHI-Y measures the frequency of the most common NSSI behaviors. The primary outcome will be the proportion of treatment remission. Remission will be defined as the absence of self-injury the past 30 days. Clinician-rated.
Internet Intervention Patient Adherence Scale (iiPAS) | Treatment week 3 and post-treatment (week 12)
  The IIPAS measures patient adherence to guided internet-delivered behavioral interventions. This scale has 5 items, and a total score ranging from 0 to 20, where 0 indicates no adherence and 20 perfect adherence. Clinician-rated.
Credibility/Expectancy Questionnaire (CEQ) - 1 item version | Treatment week 3
  CEQ measures treatment credibility and expectancy. This version of the scale has 1 item ranging from 0 to 100, with higher scores indicating greater credibility/expectancy. Self-rated (adolescent).
The Client Satisfaction Questionnaire (CSQ) | Post-treatment (week 12)
  The CSQ measures satisfaction with treatment. This scale has 8 items and a summary score ranging from 8 to 32, with higher scores indicating greater treatment satisfaction. Self-rated (adolescent and parent).
Therapist time | Post-treatment (week 12)
  Clinicians report time spent on treatment.
Number of completed sessions and modules | Post-treatment (week 12)
  Clinicians report number of completed sessions and modules for adolescents and parents.
Rate of treatment adaptions | Post-treatment (week 12)
  Clinicians report presence or absence of possible treatment adaptions (e.g., changes in therapist contact or what material to focus on).
Degree of partcipation in data collection | One-month post-treatment
  The proportion of adolescents completing the primary clinical outcome, Deliberate Self-harm Inventory - Youth version, either through interview or self-report questionnaire at one-month post-treatment
Adapted ICBT Therapist Rating Scale (ICBT-TRS) | Through study completion, an average of 1 year
  Therapist behaviors are rated separately as 0 (absence of behavior), 1 (inadequate performance), or 2 (competent). Rated by experienced clinical supervisors.

SECONDARY OUTCOMES:
Deliberate Self-harm Inventory - Youth version (DSHI-Y) | Baseline, one-, three- and twelve-months post-treatment
  The DSHI-Y measures the frequency of the most common NSSI behaviors. Change in NSSI frequency from baseline to respective follow-up will be a secondary outcome. Clinician-rated.
Children's Global Assessment Scale (CGAS) | Baseline, one-, three- and twelve-months post-treatment
  The CGAS measures global functioning on a single item ranging from 1 to 100, with a higher value indicating better functioning. Clinician-rated.
Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) | Baseline, one-, three- and twelve-months post-treatment
  The DERS-16 measures difficulties in emotion regulation. The total score ranges from 16 to 80, with higher scores indicating greater difficulties. Self-rated (adolescent and parent).
Child Health Utility 9D (CHU-9D) | Baseline, one-, three- and twelve-months post-treatment
  The CHU-9D measures health related quality of life. The scale has 9 items with a summary score between 9 and 45, where a higher score indicates greater health-related quality of life. Self-rated (adolescent).
Borderline symtom checklist supplement (BSL) | Baseline, one-, three- and twelve-months post-treatment
  The BSL supplement measures the frequency of eleven self-destructive behaviors. The total score ranges from 0 to 44 where a higher score indicates greater frequency of self-destructive behaviors. Self-rated (adolescent).
The Revised Child Anxiety and Depression Scale-Short Version (RCADS-25) | Baseline, one-, three- and twelve-months post-treatment
  The RCADS-25 measures symptoms of depression and anxiety in children and adolescents. This version has 25 items with a total score between 0 and 75, with higher scores indicating greater levels of symptoms. Self-rated (adolescent).
The Coping with Children's Negative Emotions Scale Adolescent Version (CCNES-A) | Baseline, one-, three- and twelve-months post-treatment
  The CCNES-A measures parental coping in response to adolescents' negative emotions. The CCNES-A consists of nine hypothetical scenarios accompanied by six types of responses (i.e., emotion focused, problem-focused, minimization, punitive, expressive encouragement, and distress responses). Separate summary scores are calculated per subscale (type of response) and ranges from 1 to 7, with higher scores indicating greater usage of a certain parental coping style. Self-rated (parent).
The Work and Social Adjustment Scale -Youth version (WSAS-Y) | Baseline, one-, three- and twelve-months post-treatment
  The WSAS-Y measures functional impairment in school, everyday life, friends and social life, recreation and hobbies, and family and close relationships.This 5-item scale generates a summary score between 0 and 40, with higher scores indicating greater impairment. Youths rate their own impairment. Self-rated.
The Work and Social Adjustment Scale - Parent version (WSAS-P) | Baseline, one-, three- and twelve-months post-treatment
  The WSAS-P measures functional impairment in school, everyday life, friends and social life, recreation and hobbies, and family and close relationships.This 5-item scale generates a summary score between 0 and 40, with higher scores indicating greater impairment. Parents rate their youth's impairment. Self-rated.

OTHER OUTCOMES:
Participant-rated adherence | Treatment week 3
  Two items asking the participant to rate their own adherence the past week. Self-rated (adolescent).
Credibility | Treatment week 3
  Two items asking the participant to rate change in treatment credibility from the previous treatment week. Self-rated (adolescent).
Adverse events | Post-treatment (week 12)
  A scale were participants are asked to report, describe, and rate the discomfort/impact of any negative effects or adverse events caused by their participation in the treatment. Participants rate the impact of potential adverse events when it happened and today on a scale from 1 to 4, where a higher score indicates greater impact. Self-rated (adolescent and parent).
Concomitant treatment | Post-treatment (week 12), one- and three-months post-treatment
  Participants report presence, type, focus, and change an of any potential other concomitant treatment during the trial. Self-rated (adolescent and parent).
The clinician's satisfaction with treatment adaptions | Post-treatment (week 12)
  Clinicians report their own level of satisfaction with the given treatment adaptions (one item).
Columbia-Suicide Severity Rating Scale (C-SSRS) - 6 item version | Baseline
  The C-SSRS - 6 item version measures the frequency and severity of suicidal ideation and behaviors. Clinician-rated.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Week 1 to 12
  Two items about suicidal behavior from the C-SSRS are used to measure suicidality during treatment. The items concern preparatory behavior and suicide attempts the past seven days. Self-rated (adolescent).
Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) | Week 1 to 12
  The DERS-16 measures difficulties in emotion regulation. The total score ranges from 16 to 80, with higher scores indicating greater difficulties. Self-rated (adolescent).
Deliberate Self-harm Inventory - Youth version (DSHI-Y) | Baseline, week one to 12, post-treatment, one-, three- and twelve-months post-treatment
  The DSHI-Y measures the frequency of the most common NSSI behaviors. Self-rated (adolescent).
Inventory of Statements About Self-injury (ISAS) | Baseline
  ISAS measures frequency, function, age of onset, experience of, and willingness to stop engaging in self-injury. There are 39 items describing common functions of self-injury. Participants are asked to rate if a certain function applies to them, by marking the statement as "Not relevant", "Partly relevant", or "Very relevant". Self-rated (adolescent).
Trimbos/iMTA questionnaire for Costs associated with Psychiatric illness (TIC-P) | Baseline, one-, three- and twelve-months post-treatment
  The TIC-P measures healthcare and societal resource use, including for example items on healthcare resource use, medications, school absenteeism, and parental productivity loss. Self-rated (parent).
Experiences of self- and assessor-rated nonsuicidal self-injury (NSSI) reports | Baseline, one- or three-months post-treatment
  Adolescents will be asked two questions about the format used to report NSSI: (1) "What was your experience of reporting NSSI in the different formats?", and in case where discrepancies occur between the two reporting formars between: (2) "Which frequency rating do you prefer?". Both questions will be administered by an assessor during a single assessment session.
Academic performance | 1-10 years post-treatment
  Grades and eligibility in primary school and upper secondary school, and highest education level. Registry data from the Swedish National Agency for Education and the Swedish longitudinal integrated database for health insurance and labour market studies (LISA).
Number of healthcare visits | 1-10 years post-treatment
  Registry data from the National Patient Register.
Prescription of psychotropics | 1-10 years post-treatment
  Registry data from the National Prescribed Drug Register.
Mental health disorders | 1-10 years post-treatment
  Registered psychiatric disorders. Registry data from the National Patient Register.
Reasons for eventual death | 1-10 years post-treatment
  Registry data from the National Cause of Death Register.
Suicide attempts | 1-10 years post-treatment
  Suicide attempts registered by the health care. Registry data from the National Patient Register and Regional Healthcare Registers.
Occupation | 1-10 years post-treatment
  Occupation, including unemployment and sick leave. Registry data from the Swedish longitudinal integrated database for health insurance and labour market studies (LISA).
The Revised Child Anxiety and Depression Scale (RCADS) | 1-10 years post-treatment
  The RCADS measures symptoms of depression and anxiety in children and adolescents. RCADS has 47 items with a total score between 0 and 141, with higher scores indicating greater levels of symptoms. Registry data from the National Quality Register for Child and Adolescent Mental Health Services (Q-BUP).
Children's Global Assessment Scale (CGAS) | 1-10 years post-treatment
  The CGAS measures global functioning on a single item ranging from 1 to 100, with a higher value indicating better functioning. Registry data from the National Quality Register for Child and Adolescent Mental Health Services (Q-BUP).
Kidscreen-10 | 1-10 years post-treatment
  The Kidscreen-10 measures quality of life through 10 items. The summary score ranges from 10 to 50 where a higher score indicates greater quality of life. Registry data from the National Quality Register for Child and Adolescent Mental Health Services (Q-BUP).

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Ojala, PhD, Principal Investigator — Karolinska Institutet; Johan Bjureberg, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The data is pseudonymized in accordance with Swedish and European Union laws and cannot be anonymized and published in an open repository. Study participants have consented to sharing their data with international researchers for meta-analyses. Aggregated data can be provided upon reasonable request on a case-by-case basis in compliance with current legislation and ethical permits